CLINICAL TRIAL: NCT02077413
Title: Muscle Injury Prevention & Rehabilitation in Military Personnel
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Florida (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: USAMRMC W81XH-11-1-0454
Record Dates: First submitted 2014-02-27; First posted 2014-03-04 (Estimated); Last update posted 2016-11-17 (Estimated); Status verified 2016-11

CONDITIONS: Muscle Injury
Keywords: muscle; eccentric exercise; T2 MRI

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Healthy Muscle Group (Active Comparator): Six subjects will be enrolled in this group. MRI measures will be performed at baseline and 48 hours post-exercise, when the largest amount of muscle damage is typically observed. They will be tested for maximum strength of the dorsiflexors and then undergo an eccentric exercise protocol for both lower legs on the Biodex with varying loads. Approximately two days after the exercise protocol, the participants will have another MRI of the lower legs to assess any change in T2 relaxation time as a construct of muscle edema/damage.
  Interventions: Procedure: Healthy Muscle Group
- Stretch-Contract Pre-rehabilitation Group (Experimental): All subjects will be tested initially with an MRI, blood work for creatine kinase levels (CK), subjective report of pain, range of motion (ROM) of the lower leg/ankle, and maximum strength of the dorsiflexors. They will also receive the "stretch-contract" protocol on one leg consisting of the following: a 5 second passive stretch of the dorsiflexors, followed immediately by a 5 second active isometric contraction of the dorsiflexors, and a 5 second rest/relaxation period. This cycle will continue for a duration of ~5 minutes.
  Interventions: Procedure: Stretch-Contract Pre-rehabilitation Group
- Stretch-Contract Control Group (Active Comparator): All subjects will be tested initially with an MRI, blood work for creatine kinase levels (CK), subjective report of pain, range of motion (ROM) of the lower leg/ankle, and maximum strength of the dorsiflexors.
  Interventions: Procedure: Stretch-Contract Control Group
- Muscle Atrophy (Experimental): These subjects will undergo MRI and strength testing at baseline and will also be assessed for CK levels, pain report, and ROM. They will then receive an eccentric loading paradigm for the dorsiflexor muscles of the involved leg using an isokinetic dynamometer with varying loads. Approximately two days after the exercise protocol, follow-up assessment of MRI, CK levels, pain report, ROM, and strength will be done.
  Interventions: Procedure: Muscle Atrophy

INTERVENTIONS:
Procedure: Healthy Muscle Group — Six subjects will be enrolled in this group. MRI measures will be performed at baseline and 48 hours post-exercise, when the largest amount of muscle damage is typically observed. They will be tested for maximum strength of the dorsiflexors and then undergo an eccentric exercise protocol for both lower legs on the Biodex with varying loads. Approximately two days after the exercise protocol, the participants will have another MRI of the lower legs to assess any change in T2 relaxation time as a construct of muscle edema/damage.
  Arms: Healthy Muscle Group
Procedure: Stretch-Contract Pre-rehabilitation Group — All subjects will be tested initially with an MRI, blood work for creatine kinase levels (CK), subjective report of pain, range of motion (ROM) of the lower leg/ankle, and maximum strength of the dorsiflexors. They will also receive the "stretch-contract" protocol on one leg consisting of the following: a 5 second passive stretch of the dorsiflexors, followed immediately by a 5 second active isometric contraction of the dorsiflexors, and a 5 second rest/relaxation period. This cycle will continue for a duration of ~5 minutes.
  Arms: Stretch-Contract Pre-rehabilitation Group
Procedure: Stretch-Contract Control Group — All subjects will be tested initially with an MRI, blood work for creatine kinase levels (CK), subjective report of pain, range of motion (ROM) of the lower leg/ankle, and maximum strength of the dorsiflexors.
  Arms: Stretch-Contract Control Group
Procedure: Muscle Atrophy — These subjects will undergo MRI and strength testing at baseline and will also be assessed for CK levels, pain report, and ROM. They will then receive an eccentric loading paradigm for the dorsiflexor muscles of the involved leg using an isokinetic dynamometer with varying loads. Approximately two days after the exercise protocol, follow-up assessment of MRI, CK levels, pain report, ROM, and strength will be done.
  Arms: Muscle Atrophy

SUMMARY:
The overall goal of this study is to establish a new pre-rehabilitation program in the prevention of muscle injury in the legs of healthy people serving in the military and injured individuals with muscle wasting following leg injuries. The specific goals include: 1) the amount of exercise that causes injury to healthy muscle in the lower leg of healthy people; 2) what is the effect of an intervention (pre-rehabilitation program) on decreasing how easily the muscle of the lower leg can be injured in healthy people; 3a) what amount of exercise causes injury to muscle that has recently been injured and is recovering and 3b) the effect of the new pre-rehabilitation program on the muscles of the lower leg when the muscle has recently been injured and is still recovering.

For the first goal, the investigators will determine how easily the muscle can get injured from a specific exercise in 6 healthy, conditioned men and women. Participants will perform different amounts of exercise with the lower leg muscles to see how easily the muscle can be damaged. Magnetic resonance imaging (MRI) will be used to estimate how much damage occurs with the different levels of exercise. For the second goal, the investigators will examine the effect of a new pre-rehabilitation program on decreasing how easily muscle gets damaged from the exercise we did in the first goal. The investigators will invite healthy people to participate in this goal. The investigators will use MRI, blood markers, and pain as ways of assessing muscle damage in 10 people who do the pre-rehabilitation program before exercising and 10 who do not do the new program. The third goal will focus on a) determining how easily muscle gets injured that has recently recovered from some trauma (5 people will participate in this part of the third goal), and b) determining how a pre-rehabilitation program decreases how easily a muscle that has just recovered from trauma gets injured from exercise (10 people will participate in this part of the third goal).

DETAILED DESCRIPTION:
A total of 26 healthy adults and 15 adults who have recently experienced muscle atrophy from conservative treatment after an orthopedic lower leg/ankle/foot injury that did not require surgery but did require immobilization will participate.

Magnetic resonance imaging (MRI) will be used to estimate how much damage occurs with the different levels of exercise. The investigators will be using a T2 MR which has been shown to be sensitive to injury of muscle damage.

There will be four groups in this protocol as outlined:

Healthy Muscle Group:

Six subjects will be enrolled in this group. MRI measures will be performed at baseline and 48 hours post-exercise, when the largest amount of muscle damage is typically observed. They will be tested for maximum strength of the dorsiflexors and then undergo an eccentric exercise protocol for both lower legs on the Biodex with varying loads. Approximately two days after the exercise protocol, the participants will have another MRI of the lower legs to assess any change in T2 relaxation time as a construct of muscle edema/damage.

Stretch-Contract Pre-rehabilitation Group All subjects will be tested initially with an MRI, blood work for creatine kinase levels (CK), subjective report of pain, range of motion (ROM) of the lower leg/ankle, and maximum strength of the dorsiflexors. They will also receive the "stretch-contract" protocol on one leg consisting of the following: a 5 second passive stretch of the dorsiflexors, followed immediately by a 5 second active isometric contraction of the dorsiflexors, and a 5 second rest/relaxation period. This cycle will continue for a duration of ~5 minutes.

Stretch-Contract Control Group All subjects will be tested initially with an MRI, blood work for creatine kinase levels (CK), subjective report of pain, range of motion (ROM) of the lower leg/ankle, and maximum strength of the dorsiflexors. This group will not receive the "stretch-contract" protocol.

Muscle Atrophy These subjects will undergo MRI and strength testing at baseline and will also be assessed for CK levels, pain report, and ROM. They will then receive an eccentric loading paradigm for the dorsiflexor muscles of the involved leg using an isokinetic dynamometer with varying loads.

All exercise testing will be performed on an isokinetic dynamometer by a physical therapist who has received extensive training for this piece of exercise equipment.

ELIGIBILITY:
Inclusion Criteria:

Inclusion criteria for control subjects [primary target being Reserve Officer Training Corps (ROTC) personnel]: 1) healthy individuals ages 18-40 years; and 2) ankle range of motion for the leg to be tested from 0 degrees of plantarflexion to 30 degrees of plantarflexion.

Exclusion criteria for control subjects (primary target being ROTC personnel): 1) previous history of trauma and/or surgery to the lower extremities that may limit function; 2) neurological, vascular, or cardiac problems that may limit function; 3) diabetes; 4) previous traumatic head injury or post-traumatic stress disorder; 5) a contraindication to MRI e.g.: pacemakers, metal implants which are not MRI compatible, pregnancy, and severe claustrophobia; and 6) currently performing an exercise program that specifically targets the dorsiflexor muscles.

Inclusion criteria for subjects with muscle atrophy: 1) individuals ages 18-40 years with an injury to the lower leg requiring immobilization but no surgical intervention; and 2) ankle range of motion for the leg to be tested from 0 degrees of plantarflexion to 30 degrees of plantarflexion.

Exclusion criteria for subjects with muscle atrophy: 1) previous history of trauma and/or surgery to the lower extremities, other than the injury for being immobilized, that may limit function; 2) neurological, vascular, or cardiac problems that may limit function; 3) orthopedic conditions affecting the contralateral, uninvolved lower extremity that may limit function; 4) diabetes; 5) previous traumatic head injury or post-traumatic stress disorder; and 6) a contraindication to MRI e.g.: pacemakers, metal implants which are not MRI compatible, pregnancy, and severe claustrophobia.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 41 (Actual)
Dates: Start 2014-03; Primary Completion 2016-11 (Actual); Study Completion 2016-11 (Actual)

PRIMARY OUTCOMES:
Change from Baseline in T2 relaxation time of skeletal muscle in the lower leg | Change in baseline to 48 hours
  T2 weighted spin-echo magnetic resonance imaging (MRI) will be acquired with a fixed bandwidth, a TR=3s, optimized field of view (FOV_, 7mm slice thickness, and TEs of 20, 40, 60, 80, and 100 msec. A pixel-by-pixel T2 map will be created for each slice by fitting the decay in image signal intensity (SI) to a single exponential (SI=Aexp-TE/T2+B; A=proton density) with respect to echo time (TE).
Change from Baseline in T2 relaxation time of skeletal muscle in the lower leg | Change in baseline to week 1
  T2 weighted spin-echo magnetic resonance imaging (MRI) will be acquired with a fixed bandwidth, a TR=3s, optimized field of view (FOV_, 7mm slice thickness, and TEs of 20, 40, 60, 80, and 100 msec. A pixel-by-pixel T2 map will be created for each slice by fitting the decay in image signal intensity (SI) to a single exponential (SI=Aexp-TE/T2+B; A=proton density) with respect to echo time (TE).

SECONDARY OUTCOMES:
Change from Baseline in Creatine Kinase levels | Change in baseline to 48 hours
  Approximately 10 ml of blood will be analyzed for CK levels.
Change from Baseline in Muscle water proton T2 | Change in baseline to 48 hours
  A spectroscopic relaxometry sequence may be implemented to quantify changes in muscle water proton (1H2O) T2. Sixteen echoes may be acquired in the musculature of the lower leg under fully relaxed conditions (TR=9 s). This sequence will allow for both the determination of global T2 as well as multiexponential fitting of the T2 decay using non-negative least squares analysis.
Change from Baseline in Muscle contractile area | Change in baseline to 48 hours
  A T1 weighted MRI will be used to measure changes in muscle contractile area. Using a coronal localizer scout, transaxial images (~50 slices) will be acquired along the length of the muscles, oriented perpendicular to the long bone (tibia or femur). All images may be acquired with optimized FOV(~12x12 cm2), TR=17 ms, TE=2ms, Number of Excitations (NEX)=2, and a flip angle of 20˚. Images may be acquired with an encoding matrix of 256x256 and 3mm slice thickness.
Change from Baseline in Isometric muscle strength of the ankle dorsiflexors | Change in baseline to 48 hours
  Ankle dorsiflexor muscles will be tested using an isokinetic dynamometer. The measurement of the peak isometric torque will be taken with the subjects seated in an upright position using a standardized set-up. Assessment of the dorsiflexors will be performed with the ankle in slight plantarflexion and the knee in slight flexion. The subjects will have three to ten maximal trials of ~5 sec which will be performed and the peak torque recorded. A rest time of ~1 minute will be provided between each contraction. A visual feedback display will be used to motivate the subjects to reach their maximum torque output. Peak torque measures may be normalized to maximal cross-sectional area (CSAmax) to assess muscle specific torque.
Change from Baseline in Pain scores on a visual analog scale | Change in baseline to 48 hours
  Subjects who participate in pain assessment will be asked to rate any pain they are experiencing at the time of assessment using a numeric rating scale of a line anchored at 0 (no pain sensation at all) and 100 (worst pain imaginable). Subjects will be asked to rate any pain by making a mark on the 100 mm line.
Change from Baseline in ankle Range of Motion (ROM) | Change in baseline to 48 hours
  Subjects who participate in ROM testing will be positioned supine with their knee fully extended, and ankle ROM for both dorsiflexion and plantarflexion will be determined actively with a standard goniometer.
Change from Baseline in Creatine Kinase levels | Change in baseline to week 1
  Approximately 10 ml of blood will be analyzed for CK levels.
Change from Baseline in Muscle water proton T2 | Change in baseline to week 1
  A spectroscopic relaxometry sequence may be implemented to quantify changes in muscle water proton (1H2O) T2. Sixteen echoes may be acquired in the musculature of the lower leg under fully relaxed conditions (TR=9 s). This sequence will allow for both the determination of global T2 as well as multiexponential fitting of the T2 decay using non-negative least squares analysis.
Change from Baseline in Muscle contractile area | Change in baseline to week 1
  A T1 weighted MRI will be used to measure changes in muscle contractile area. Using a coronal localizer scout, transaxial images (~50 slices) will be acquired along the length of the muscles, oriented perpendicular to the long bone (tibia or femur). All images may be acquired with optimized FOV(~12x12 cm2), TR=17 ms, TE=2ms, Number of Excitations (NEX)=2, and a flip angle of 20˚. Images may be acquired with an encoding matrix of 256x256 and 3mm slice thickness.
Change from Baseline in Isometric muscle strength of the ankle dorsiflexors | Change in baseline to week 1
  Ankle dorsiflexor muscles will be tested using an isokinetic dynamometer. The measurement of the peak isometric torque will be taken with the subjects seated in an upright position using a standardized set-up. Assessment of the dorsiflexors will be performed with the ankle in slight plantarflexion and the knee in slight flexion. The subjects will have three to ten maximal trials of ~5 sec which will be performed and the peak torque recorded. A rest time of ~1 minute will be provided between each contraction. A visual feedback display will be used to motivate the subjects to reach their maximum torque output. Peak torque measures may be normalized to maximal cross-sectional area (CSAmax) to assess muscle specific torque.
Change from Baseline in Pain scores on a visual analog scale | Change in baseline to week 1
  Subjects who participate in pain assessment will be asked to rate any pain they are experiencing at the time of assessment using a numeric rating scale of a line anchored at 0 (no pain sensation at all) and 100 (worst pain imaginable). Subjects will be asked to rate any pain by making a mark on the 100 mm line.
Change from Baseline in ankle Range of Motion (ROM) | Change in baseline to week 1
  Subjects who participate in ROM testing will be positioned supine with their knee fully extended, and ankle ROM for both dorsiflexion and plantarflexion will be determined actively with a standard goniometer.

CONTACTS AND LOCATIONS:
Overall Officials: Donovan J Lott, PT, PhD, Principal Investigator — University of Florida
Locations (1):
- University of Florida, Gainesville, Florida, United States